CLINICAL TRIAL: NCT04413214
Title: Safety and Efficacy Evaluation of Carrimycin in Patients With Locally Advanced, Recurrent, or Metastatic Head and Neck Squamous Cell Carcinoma (Non NPC): A Phase I Trial
Brief Title: Carrimycin in Patients With Locally Advanced, Recurrent, or Metastatic HNSCC (Non NPC): A Phase I Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clarion I
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2021-12

CONDITIONS: Oral Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — carrimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Group (Experimental): The 3x3 dose escalation design will be adopted, including 200mg, 400mg and 600mg of Carrimycin; and three subjects at each dose level initially. If there is no DLT in the dose level of 200mg, the dose level of 400mg will be followed; if there is one DLT in the dose level of 200mg, another three patients will be added in the dose level of 200mg; if there is no DLT occurs in the another three patients, the dose level of 400mg will also be followed; if there is one DLT in the another three patients, the trial will be closed. The same condition to the dose level of 400mg and 600mg.
  Interventions: Drug: Carrimycin

INTERVENTIONS:
Drug: Carrimycin — The study involves three dose groups: 200mg, 400mg and 600mg. Three patients are planned for each dose group. Starting from the low dose group, the treatment to three patients in the 200mg dose group: 200mg of Carrimycin after meals every morning (po) for three weeks, and then discontinue for one week, the tolerance and efficacy evaluation will be performed after the 4 weeks. DLT will be recorded during the 4 weeks.

SUMMARY:
The trial is a study conducted to evaluate the safety, tolerability and PK characteristics of Carrimycin tablet and measure its anti-tumor efficacy initially in the treatment of patients with locally advanced, recurrent, or metastatic head and neck squamous cell carcinoma (non NPC).

DETAILED DESCRIPTION:
This study is a prospective open phase-I study to investigate the safety, tolerability and PK characteristics of Carrimycin tablet in the treatment of patients with locally advanced, recurrent, or metastatic head and neck squamous cell carcinoma (non NPC). The 3x3 dose escalation design will be adopted, including 200mg, 400mg and 600mg of Carrimycin; and three subjects at each dose level initially. If there is no DLT in the dose level of 200mg, the dose level of 400mg will be followed; if there is one DLT in the dose level of 200mg, another three patients will be added in the dose level of 200mg; if there is no DLT occurs in the another three patients, the dose level of 400mg will also be followed; if there is one DLT in the another three patients, the trial will be closed. The same condition to the dose level of 400mg and 600mg. If a patient fails to receive the full prescribed dose for reasons other than DLT at the time of the first administration, the patient will be replaced. Carrimycin treatment to the patients with DLT will be discontinued immediately and they will enter the follow-up period and will not be replaced. The study consists of screening period, treatment period and follow-up period. The treatment period continues until the patients develop progressive disease, dies, lost to follow-up or withdraw informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, recurrent, or metastatic head and neck squamous cell carcinoma (non NPC) confirmed by histopathological or cytological diagnosis
* Expected life expectancy is no less than 6 months;
* ECOG PS is 0, 1 or 2;
* Subjects should be enrolled at least 4 weeks after the lastest treatment of surgery, radiotherapy, chemotherapy, or biotherapy, etc.
* The laboratory inspection indexes should meet the following requirements: Leukocyte>3×109/L, Neutrophils>1.5×109/L, Platelet count>75×109/L，Hemoglobin>80g/L, Serum total bilirubin<1.5ULN, ALT or AST<2.5ULN, Creatinine<2.0ULN, BUN<2.0ULN, Maximum extension of APTT normal is within 10s, Maximum extension of PT normal is within 3s.
* Women of reproductive age (18-45 years) must have a negative urine pregnancy test and agree to receive effective contraception. Male subjects must voluntarily receive appropriate contraception.

Exclusion Criteria:

* There is still any undiminished CTCAE grade 2 or higher toxicity from previous anti-cancer treatments;
* There are significant cardiovascular abnormalities (e.g. myocardial infarction, upper-cavity venous syndrome, heart disease of grade 2 or higher diagnosed according to the New York Heart Association (NYHA) classification criteria 3 months prior to enrollment);
* There is active severe clinical infection (>NCI-CTCAE V5.0 Level 2)
* Urine routine shows albuminuria ≥ ++, but if albuminuria at baseline ≥ ++, patients with albuminuria /24h<1g measured quantitatively based on 24-hour urine collection can be enrolled;
* Allergic to macrolides;
* Uncontrolled hypertension (systolic > 150 mmHg and / or diastolic >100mmHg) or clinically significant (e.g. active) cardiovascular diseases - such as stroke (≤ 6 months before randomization), myocardial infarction (≤ 6 months before randomization), unstable angina pectoris, congestive heart failure of New York Heart Association (NYHA) functional class III or above, or serious arrhythmia that cannot be controlled with drugs or has potential impact on trial treatment.
* Known to have acute or chronic active HBV or HCV infection and need antiviral treatment with non nucleoside drugs;
* Women pregnant or lactation;
* Having participated in other clinical studies and received any other investigational drug for treatment within 30 days before enrollment;
* Having taken macrolide antibiotics (azithromycin, erythromycin, roxithromycin, clarithromycin, dirithromycin, spiramycin, acetylspiramycin, midecamycin, rokitamycin, meleumycin, josamycin, leucomycin, miocamycin) within 3 days before enrollment;
* Other cases considered inappropriate by the investigator to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Two years
  According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) 5.0, evaluate adverse events occurred during the whole study period.
Dose limiting toxicity | Four weeks
  According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) 5.0, observe the dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Objective response rate to Carrimycin | Four weeks
  Including complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD)
Progression-free survival | Two years
  The period between the time a patient with a cancer disease begins to receive treatment and observe the disease progression or die for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Lai-ping Zhong, PhD/MD, Principal Investigator — Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ninth People's Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No